CLINICAL TRIAL: NCT04833647
Title: Influence of Prematurity and Its Respiratory Sequel on Exercise Testing in Childhood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ori Hochwald , MD, Director, NICU, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0239-14-RMB
Record Dates: First submitted 2021-04-03; First posted 2021-04-06 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: The Peak Oxygen Consumption (VO2max) Was Measured and Served as the Primary Endpoint of the Study

STUDY DESIGN:
Intervention Model Description: Participants performed CPET on an electronically braked cycle ergometer . During the exercise testing, serial saturation, heart rate and blood pressure measurements were obtained. The peak oxygen consumption (VO2max) was measured and served as the primary endpoint of the study. A CPET technician and a senior pediatrician were present and monitored the participants' condition during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Term (Other): 7-10 years old born at 37-42 weeks gestation
  Interventions: Diagnostic Test: Cardio-Pulmonary-Exercise-Testing (CPET)
- Late preterms (Other): 7-10 years old born at 34.0-36.6 weeks gestation
  Interventions: Diagnostic Test: Cardio-Pulmonary-Exercise-Testing (CPET)
- Preterms with BPD (Other): 7-10 years old born before 30 weeks gestation with the diagnosis of BPD: the need for oxygen at 36 weeks gestation and/or flow or 3LPM or more, and/or the need for CPAP or invasive ventilation
  Interventions: Diagnostic Test: Cardio-Pulmonary-Exercise-Testing (CPET)
- pretermas without BPD (Other): 7-10 years old born before 30 weeks gestation without the diagnosis of BPD (without the need for oxygen at 36 weeks gestation and/or flow or 3LPM or more, and/or the need for CPAP or invasive ventilation)
  Interventions: Diagnostic Test: Cardio-Pulmonary-Exercise-Testing (CPET)

INTERVENTIONS:
Diagnostic Test: Cardio-Pulmonary-Exercise-Testing (CPET) — Cardio-Pulmonary-Exercise-Testing (CPET) . During the exercise testing, serial saturation, heart rate and blood pressure measurements were obtained. The peak oxygen consumption (VO2max) was measured and served as the primary endpoint of the study

SUMMARY:
Prospective study comparing hemodynamic and respiratory changes and exercise capacity during Cardio-Pulmonary-Exercise-Testing (CPET) in 4 groups of infants; Three different groups of premature infants and term controls

DETAILED DESCRIPTION:
The study population included 4 groups of infants; preterm infants born < 300 weeks' gestation with BPD (i.e. oxygen dependence for at least 28 postnatal days 5), preterm infants born < 300 weeks' gestation without BPD, late preterm infants (born at 340-366 weeks' gestation) and term controls.

Pulmonary function testing and spirometry were measured Participants performed CPET on an electronically braked cycle ergometer. During the exercise testing, serial saturation, heart rate and blood pressure measurements were obtained.

The peak oxygen consumption (VO2max) was measured and served as the primary endpoint of the study.

ELIGIBILITY:
Inclusion Criteria:

* 7-10 years of age
* The ability to ride stationary bicycles as assessed by the parents.

Exclusion Criteria:

* Immobility
* An acute febrile or upper respiratory illness in the last 2 weeks
* The use systemic or inhaled steroids or antiepileptic drugs in the previous month
* Inhaled bronchodilator use in the previous 24 hours
* A chronic lung illness (with the exception of BPD and asthma)
* Congenital cardiac defect (with the exception of atrial septal defect and patent foramen ovale).

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
The peak oxygen consumption (VO2max) | During the 1 day test
  The peak oxygen consumption (VO2max)

IPD SHARING:
Plan to Share IPD: Undecided